CLINICAL TRIAL: NCT04724551
Title: The Neutrophil-to-Lymphocyte Ratio at Post-operative Day 3: a Simple Tool to Exclude Clinically Relevant Postoperative Pancreatic Fistula After Pancreatoduodenectomy
Brief Title: The Neutrophil-to-Lymphocyte Ratio to Exclude Pancreatic Fistula
Acronym: NLR
Status: Completed | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: NLR-IPC 2020-058
Record Dates: First submitted 2021-01-19; First posted 2021-01-26 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-01

CONDITIONS: Pancreas Neoplasm
Keywords: Pancreatic fistula; Neutrophil-to-Lymphocyte Ratio; Pancreatoduodenectomy
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Fistula | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: pancreatoduodenectomy (PD) — A pancreaticogastrostomy or -jejunostomy duct-to-mucosa was achieved according to the surgeon's preference and pancreatic texture.

SUMMARY:
There is still no consensus on whether drain fluid amylase (DFA) level, C-reactive protein (CRP) level, or complex scores predict clinically relevant postoperative pancreatic fistula (CR-POPF). The aim of this study is to determine the accuracy of simple biochemical parameters (leucocytes, neutrophils, lymphocytes, Neutrophil to Lymphocytes Ratio (NLR), at postoperative days 1 and 3) to exclude the diagnosis of CR-POPF.

DETAILED DESCRIPTION:
From January 1, 2012 to December 31, 2020, consecutive patients underwent PD performed at Institut Paoli-Calmettes for various pathologies. Data were entered prospectively into a clinical database (NCT02871336).

The cohort was split into 3 groups:

* a training cohort ;
* an internal validation cohort (Paoli Calmettes institute);
* an external validation cohort (Rennes Pontchaillou Hospital).

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent pancreatoduodenectomy

Exclusion Criteria:

* Total pancreatectomy
* Enucleation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 3 cohorts, which were as follows: the set of 451 patients was randomly sampled following a ratio 2:1 into a training (n=301) and a validation (n=150) cohort to respectively determine and validate the accuracy, best timing, and cut-off for the surrogate markers, then validated in an external cohort (n=197).
Sampling Method: Probability Sample
Enrollment: 648 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of clinically relevant pancreatic fistula | at hospital discharge assessed up to 30 days
  Clinically relevant postoperative pancreatic fistula according to the 2016 International Study Group of Pancreatic Surgery definition

SECONDARY OUTCOMES:
Biological markers | Postoperative day one and three
  Identification of biological markers to exclude clinically relevant postoperative pancreatic fistula

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Turrini, PD, Principal Investigator — Institut Paoli-Calmettes- (IPC)

IPD SHARING:
Plan to Share IPD: No